CLINICAL TRIAL: NCT06315296
Title: Txt4fasting: An Interactive Mobile Time-Restricted Eating Diet Intervention for Patients With Brain Metastases to Maximize Radiation Outcomes
Brief Title: An Interactive Time-Restricted Diet Intervention (txt4fasting) for Reducing Neurocognitive Decline and Improving Survival in Patients With Brain Metastases From Breast or Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: iRISID-2023-1985; JT 31844 (Other: JeffTrial Number)
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Breast Carcinoma; Metastatic Lung Carcinoma; Metastatic Malignant Neoplasm in the Brain; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Brain Neoplasms | interventions — Nutrition Assessment; Radiosurgery; Specimen Handling; Magnetic Resonance Spectroscopy; X-Rays; Mental Status and Dementia Tests; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (txt4fasting) (Experimental): Patients follow a time-restricted diet, receive interactive positive reinforcement messages, and record food intake using the txt4fasting platform daily for 30 days. Patients receive counseling calls twice weekly in weeks 1 and 2 then once weekly in weeks 3 and 4. Patients then undergo SRS on study. Patients also undergo blood sample collection and brain MRI throughout study.
  Interventions: Behavioral: Behavioral Dietary Intervention; Other: Text Message-Based Navigation Intervention; Other: Internet-Based Intervention; Behavioral: Dietary Counseling and Surveillance; Radiation: Stereotactic Radiosurgery; Procedure: Biospecimen Collection; Procedure: Magnetic Resonance Imaging; Other: Neurocognitive Assessment; Other: Questionnaire Administration; Other: Interview
- Arm II (attention control) (Active Comparator): Patients receive text messages about healthy eating habits and food suggestions twice daily and record food intake using txt4fasting program for 30 days. Patients then undergo SRS on study. Patients also undergo blood sample collection and brain MRI throughout study.
  Interventions: Other: Internet-Based Intervention; Radiation: Stereotactic Radiosurgery; Other: Text Message-Based Navigation Intervention; Procedure: Biospecimen Collection; Procedure: Magnetic Resonance Imaging; Other: Neurocognitive Assessment; Other: Questionnaire Administration; Other: Interview

INTERVENTIONS:
Behavioral: Behavioral Dietary Intervention — Follow a time-restricted diet
  Arms: Arm I (txt4fasting)
Other: Text Message-Based Navigation Intervention — Receive interactive positive reinforcement messages
  Other Names: Automated Text Message-Based Navigation; Text Message-Based Navigation
  Arms: Arm I (txt4fasting)
Other: Internet-Based Intervention — Use txt4fasting platform
  Arms: Arm I (txt4fasting)
Behavioral: Dietary Counseling and Surveillance — Receive counseling calls
  Arms: Arm I (txt4fasting)
Radiation: Stereotactic Radiosurgery — Undergo SRS
  Other Names: SRS; Stereotactic External Beam Irradiation; stereotactic external-beam radiation therapy; stereotactic radiation therapy; Stereotactic Radiotherapy; stereotaxic radiation therapy; stereotaxic radiosurgery
  Arms: Arm I (txt4fasting)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
  Arms: Arm I (txt4fasting)
Procedure: Magnetic Resonance Imaging — Undergo brain MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging; Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; nuclear magnetic resonance imaging; sMRI; Structural MRI
  Arms: Arm I (txt4fasting)
Other: Neurocognitive Assessment — Ancillary studies
  Arms: Arm I (txt4fasting)
Other: Questionnaire Administration — Ancillary studies
  Arms: Arm I (txt4fasting)
Other: Interview — Ancillary studies
  Arms: Arm I (txt4fasting)
Other: Internet-Based Intervention — Use txt4fasting platform
  Arms: Arm II (attention control)
Radiation: Stereotactic Radiosurgery — Undergo SRS
  Other Names: SRS; Stereotactic External Beam Irradiation; stereotactic external-beam radiation therapy; stereotactic radiation therapy; Stereotactic Radiotherapy; stereotaxic radiation therapy; stereotaxic radiosurgery
  Arms: Arm II (attention control)
Other: Text Message-Based Navigation Intervention — Receive text messages about healthy eating habits and food suggestions
  Other Names: Automated Text Message-Based Navigation; Text Message-Based Navigation
  Arms: Arm II (attention control)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
  Arms: Arm II (attention control)
Procedure: Magnetic Resonance Imaging — Undergo brain MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging; Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; nuclear magnetic resonance imaging; sMRI; Structural MRI
  Arms: Arm II (attention control)
Other: Neurocognitive Assessment — Ancillary studies
  Arms: Arm II (attention control)
Other: Questionnaire Administration — Ancillary studies
  Arms: Arm II (attention control)
Other: Interview — Ancillary studies
  Arms: Arm II (attention control)

SUMMARY:
This clinical trial tests the effectiveness of an interactive time-restricted diet intervention (txt4fasting) in reducing neurocognitive decline and improving survival outcomes after stereotactic radiosurgery in patients with breast or lung cancer that has spread to the brain (brain metastases). Lung cancer and breast cancer are the two most frequent causes of brain metastases. The diagnosis of brain metastases is associated with poorer survival and tumor-induced and treatment-related side effects. Stereotactic radiosurgery is a type of external radiation therapy that uses special equipment to position the patient and precisely give a single large dose of radiation to a tumor. Patients who receive stereotactic radiosurgery for brain metastases may experience less neurocognitive side effects than with other types of brain radiation, but may still be at risk for their brain metastases growing, spreading, or getting worse. Patients with obesity and diabetes have been shown to have worse survival and increased radiation-related side effects. Evidence demonstrates that simply changing meal timing can have a positive impact on multiple health outcomes. Time-restricted eating, or prolonged nighttime fasting, has been proven to have positive effects on heart disease risk reduction, weight control management and chemotherapy side effect reduction. Txt4fasting may be effective in decreasing neurocognitive decline and improving survival outcomes in patients undergoing stereotactic radiosurgery for brain metastases from breast or lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To examine the feasibility and acceptability of the txt4fasting intervention.

SECONDARY OBJECTIVES:

I. To compare neurocognitive function decline between the intervention and the control arms.

II. To compare progression free survival (PFS) between the intervention and the control arms.

TERTIARY (EXPLORATORY) OBJECTIVE:

I. To evaluate the change in biomarkers, from baseline to the end of the study, between the intervention and the control arms.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients follow a time-restricted diet, receive interactive positive reinforcement messages, and record food intake using the txt4fasting platform daily for 30 days. Patients receive counseling calls twice weekly in weeks 1 and 2 then once weekly in weeks 3 and 4. Patients then undergo stereostactic radiosurgery (SRS) on study. Patients also undergo blood sample collection and brain magnetic resonance imaging (MRI) throughout study.

ARM II: Patients receive text messages about healthy eating habits and food suggestions twice daily and record food intake using txt4fasting program for 30 days. Patients then undergo SRS on study. Patients also undergo blood sample collection and brain MRI throughout study.

After completion of study intervention, patients are followed up immediately at the end of the intervention, and at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Pathologically proven breast or lung cancer primary malignancy confirmed
* Body mass index (BMI) ≥ 25 kg/m^2
* SRS candidate (1-10 MRI detected brain metastases as per the discretion of radiologist) as determined by the treating physician
* Chemotherapy, hormone, and immune therapy will be allowed concurrently
* Willing and able to comply with the protocol for the duration of the study
* Able to speak, read and write English
* Negative pregnancy test if childbearing potential
* Owns a mobile phone with mobile text messaging (TXT) capability

Exclusion Criteria:

* Inability to tolerate a normal diet (may include an active malabsorption syndrome at the time of consent [i.e. Crohn's disease, major bowel resection leading to permanent malabsorption])
* Not a SRS candidate as determined by the treating physician
* Prior brain surgery ≤ 14 days prior to enrollment
* Intractable seizures while on adequate anticonvulsant therapy-more than 1 seizure per week for the past 2 months
* Patient with a diagnosis of glioma, or other World Health Organization (WHO) grade II-IV primary brain tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Accrual rate | Up to 5 years
  Feasibility will be defined as 70% of eligible patients reached consent and enroll. Accrual rate will be summarized using percentage and 95% exact confidence intervals.
Attrition rate | Up to 6 months post intervention
  Feasibility will be defined as 70% of enrolled participants complete post-intervention follow-up. Attrition rate will be summarized using percentage and 95% exact confidence intervals.
Time-restricted eating (TRE) compliance rate | Up to 6 months post intervention
  Feasibility will be defined as 70% of participants are compliant with 70% of the intervention days with suggested TRE. TRE compliance rate will be summarized using percentage and 95% exact confidence intervals.
Incidence of adverse effects (AEs) | Up to 6 months post intervention
  AEs will be graded for severity according to the Common Terminology Criteria for Adverse Events.
Patient satisfaction | Up to 6 months post intervention
  Acceptability will be measured through a validated treatment satisfaction measure and patient interview data. Acceptability will be established by a group median score ≥ 28 on the Coping Strategies Questionnaire-837. Patient satisfaction will be summarized using percentage and 95% exact confidence intervals.

SECONDARY OUTCOMES:
Neurocognitive function decline | At baseline
  Neurocognitive function decline will be measured on the Cambridge Neuropsychological Test Automated Battery. Each of the five endpoints will be modeled using linear mixed-effects models with the fixed effects of treatment arm and time as well as their interaction, and random effect of the subject.
Neurocognitive function decline | at the end of the 30-day intervention
  Neurocognitive function decline will be measured on the Cambridge Neuropsychological Test Automated Battery. Each of the five endpoints will be modeled using linear mixed-effects models with the fixed effects of treatment arm and time as well as their interaction, and random effect of the subject.
Neurocognitive function decline | at 3 month follow up
  Neurocognitive function decline will be measured on the Cambridge Neuropsychological Test Automated Battery. Each of the five endpoints will be modeled using linear mixed-effects models with the fixed effects of treatment arm and time as well as their interaction, and random effect of the subject.
Neurocognitive function decline | at 6 month follow up
  Neurocognitive function decline will be measured on the Cambridge Neuropsychological Test Automated Battery. Each of the five endpoints will be modeled using linear mixed-effects models with the fixed effects of treatment arm and time as well as their interaction, and random effect of the subject.
Intracranial progression free survival (PFS) | Time between SRS to progression of brain metastases, assesed up to 6 months post intervention
  Intracranial PFS of brain metastases will be detected by magnetic resonance imaging. Intracranial PFS between the two treatment groups will be compared using a two-sided log-rank test with the significance level of 0.05.

CONTACTS AND LOCATIONS:
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States